CLINICAL TRIAL: NCT05643170
Title: A Multi-center, Open-label Study to Assess the Effectiveness, Long-term Safety, Tolerability, and Durability of Effect of KarXT in Patients With DSM-5 Diagnosis of Schizophrenia
Brief Title: An Open-label Study to Assess the Long-term Safety, Tolerability, Effectiveness, and Durability of Effect of KarXT in Patients With DSM-5 Diagnosis of Schizophrenia
Acronym: PENNANT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company's business decision.
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAR-014
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — KarXT 50 mg/20 mg BID KarXT 100mg/20 mg BID KarXT 125mg/30 mg BID

SUMMARY:
This is a Phase 3b, 3-year, open-label, multi-center study in which patients with DSM-5 diagnosis of schizophrenia whose current medication(s) is not well tolerated and/or clinical symptoms are not well controlled will be switched to receive KarXT.

The primary objectives of the study are to assess the long-term safety and tolerability of KarXT and assess effectiveness, persistence, and durability of effect of KarXT through the Investigator Assessment Questionnaire (IAQ) and Clinical Global Impression - Severity of Illness (CGI-S) scale in patients with a diagnosis of schizophrenia.

The secondary objectives are to further assess the effectiveness using the Clinical Global Impression, Global Improvement (CGI-I), long-term safety and tolerability of KarXT, and evaluation of scores from multiple additional patient scales and assessments throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is aged 18 to 65 years, inclusive, at screening.
2. Patient can provide informed consent.

   1. A signed informed consent form (ICF) must be provided before any study assessments are performed.
   2. Patient must be fluent (oral and written) in the language of the ICF to consent.
3. Patient has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM 5 (American Psychiatric Association, 2013) criteria and has been in the continuous care of the clinician or practice for at least 6 months prior to entering the study.
4. The patient is dissatisfied with the side effects or general tolerability of their current antipsychotic medication, and for this reason, desires to change medications. Or, the patient is dissatisfied with the overall effectiveness or benefit of their current antipsychotic medication, and for this reason, desires to change medications.
5. The patient has not required psychiatric hospitalization, acute crisis intervention, or other increase in their level of care due to symptom exacerbation within 4 weeks of screening, and in the opinion of the investigator, is psychiatrically stable to be managed in an outpatient setting.
6. The patient has a CGI-S score of ≤4 (moderately severe or less) at screening and baseline visits.
7. For at least 30 days prior to screening, the patient must have been prescribed and have taken an oral antipsychotic medication daily at a dose and frequency consistent with the drug label.
8. Patient has an identified, reliable caregiver/informant that is willing (by informed consent) and able to respond to the ZBI 22 caregiver burden scale at specified visits. If the patient has been the patient of the investigator for ≥6 months and, in the opinion of the investigator, the patient is self-sufficient, then a caregiver/informant may not be necessary.
9. Patient resides in a stable living situation and is anticipated to remain in a stable living situation for the duration of the study, in the opinion of the investigator.
10. If a woman of childbearing potential (WOCBP) or a man whose sexual partner(s) is a WOCBP, the patient must be willing and able to adhere to the contraception guidelines as defined in Section 12.1 Appendix 1.

Exclusion Criteria:

1. Any primary DSM-5 disorder diagnosis other than schizophrenia within 12 months before screening. Exclusionary disorders include, but are not limited to, bipolar I or II disorder and schizoaffective disorder. Symptoms of mild mood dysphoria or anxiety are allowed, as long as these symptoms are not the primary focus of treatment.
2. The patient has a history of or presence of a clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, is likely to jeopardize the safety of the patient or the validity of the study results.
3. Patient has a history of or is at high risk of urinary retention, gastric retention, or narrow angle glaucoma.
4. Patient has a history of irritable bowel syndrome (with or without constipation) or constipation requiring treatment for more than 30 days within the last 6 months.
5. Clinically significant abnormal finding on the physical examination, medical history, electrocardiogram (ECG), or clinical laboratory results at screening.
6. Patient is pregnant, lactating, or less than 3 months postpartum.
7. Patient has tested positive for coronavirus disease 2019 (COVID-19) within 2 weeks of screening and/or baseline or patients who have prolonged symptoms of past infection, long COVID, that, in the opinion of the investigator, may interfere with the interpretation of safety during the study.
8. Patient with extreme concerns relating to global pandemics, such as COVID-19, that precludes study participation.
9. Patient is currently or recently (within 4 weeks of screening) involuntary hospitalization or incarceration.
10. Patient participated in another clinical study in which they received an experimental or investigational drug agent within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Advanced Discovery Research, LLC, Atlanta, Georgia
  - Seven Counties Services, Inc., Louisville, Kentucky
  - Mid Ohio Behavioral Health, Columbus, Ohio
  - OnSite Clinical Solutions, LLC, Rock Hill, South Carolina
  - Integrated Clinical Research, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KarXT: Participants started on a lead-in dose of KarXT 50/20 mg (xanomeline 50 mg/trospium chloride 20 mg), twice daily (BID) Day 1 to Day 7. Followed by the following titration schedule:
  * Week 1 (Days 1 to 7) - KarXT 50/20 mg, BID.
  * Week 2 (Days 8 to 14) - KarXT 100/20 mg (xanomeline 100 mg/trospium chloride 20 mg), BID or remain on 50/20 mg, BID.
  * Week 3 (Days 15 to 21) - KarXT 125/30 mg (xanomeline 125 mg/trospium chloride 30 mg), BID or 100/20 mg, BID.
  * Weeks 4 to 156 (Days 22 to 1092) - Flexible dosing based on tolerability and clinical response to KarXT 50/20 mg, KarXT 100/20 mg, and KarXT 125/30 mg, BID.
Period: Overall Study
Arm/Group | KarXT
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrew from study treatment due to study termination | 3
Not completed — Adverse event (AE) that lead to treatment discontinuation | 1

BASELINE CHARACTERISTICS:
Arm/Group | KarXT
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Discontinuation
Description: An Adverse Event (AE) is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening, worsens during the study, regardless of the suspected cause of the event.
Time Frame: From first dose to 28 days post last dose (up to approximately 113 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 4
Participants | 1

2. Primary Outcome: Investigator Assessment Questionnaire (IAQ) Scores
Description: The Investigator's Assessment Questionnaire (IAQ) evaluates all health concerns associated with antipsychotic use in patients with schizophrenia or schizoaffective disorder. The IAQ total score is defined as the sum of 10 items (positive symptoms, negative symptoms, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, EPS, cognition, energy, and mood) for a total max score of 50; each item is rated on a 5-point Likert scale (1 = Much better, 2 = Slightly better, 3 = About the same, 4 = Slightly worse, and 5 = Much worse) where higher score indicate increased health concerns.
Time Frame: At visit 1, 3, 5 (Baseline, week 4, 8), and early termination visit (study day 85)
Population: Modified Intent-to-Treat (mITT) population (All patients who are enrolled and received KarXT through week 8) with available IAQ scores at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | KarXT
Number analyzed (Participants) | 2
Score on a scale
  Visit 1 (Baseline) | 30.00 (0.000)
  Visit 3 (Week 4) | 29.50 (4.950)
  Visit 5 (Week 8) | 32.50 (2.121)
  Early Termination Visit | 31.00 (1.414)

3. Primary Outcome: Clinical Global Impression - Severity of Illness (CGI-S) Scores
Description: The Clinical Global Impression - Severity (CGI-S) is a rating scale completed independently by a clinician that is used to measure illness and symptom severity in subjects with mental disorders. It is used to rate the severity of a subject's illness at the time of assessment. The modified CGI-S asks the clinician 1 question: "Considering your total clinical experience, how mentally ill is the subject at this time?" The clinician's answer is rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects.
Time Frame: At visit 1, 2, 3, 5 (baseline, week 2, 4, 8)
Population: Modified Intent-to-Treat (mITT) population (All patients who are enrolled and received KarXT through week 8) with available CGI-S scores at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | KarXT
Number analyzed (Participants) | 2
Score on a scale
  Visit 1 (Baseline) | 3.00 (0.000)
  Visit 2 (Week 2) | 3.00 (0.000)
  Visit 3 (Week 4) | 3.00 (0.000)
  Visit 5 (Week 8) | 3.50 (0.707)

4. Secondary Outcome: The Number of Participants With Serious Treatment-Emergent Adverse Events (TESAEs)
Description: An SAE is any untoward medical occurrence that, in the view of either the investigator or Sponsor that:
  * Results in death.
  * Is life-threatening.
  * Results in inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity.
  * Is a congenital anomaly/birth defect.
  * Other important medical events
Time Frame: From first dose to 28 days post last dose (up to approximately 113 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 4
Participants | 1

5. Secondary Outcome: The Number of Participants With Treatment-Emergent Adverse Events of Special Interest (AESI)
Description: An Adverse Event (AE) is any symptom, physical sign, syndrome, or disease that either emerges during the study or, if present at Screening, worsens during the study, regardless of the suspected cause of the event. AESIs include orthostasis and liver function test (LFT) elevations (inclusive of drug induced liver injury [DILI].
  Orthostasis will be defined as the patient being symptomatic with at least one of the following differences in orthostatic vitals between sitting position and standing after 2 minutes:
  * A decrease of systolic BP of 20 mmHg or more.
  * A decrease in diastolic BP of 10 mmHg or more.
  * An increase in HR of 30 bpm or more.
Time Frame: From first dose to 28 days post last dose (up to approximately 113 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT
Number analyzed (Participants) | 4
Participants | 1

6. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Score
Description: The Clinical Global Impression - Improvement (CGI-I) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Clinicians are asked: "Compared to the patient's condition at baseline, this patient's [average] condition has...?", and they rate as: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
Time Frame: At visit 2, 3, 5 (Weeks 2, 4, 8)
Population: Modified Intent-to-Treat (mITT) population (All patients who are enrolled and received KarXT through week 8) with available CGI-I scores at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | KarXT
Number analyzed (Participants) | 2
Score on a scale
  Visit 2 (Week 2) | 3.50 (0.707)
  Visit 3 (Week 4) | 4.50 (0.707)
  Visit 5 (Week 8) | 4.50 (0.707)

7. Secondary Outcome: Medication Satisfaction Questionnaire (MSQ) Score
Description: The Medication Satisfaction Questionnaire (MSQ) is a single-item questionnaire that evaluates satisfaction with antipsychotic medication in schizophrenia patients rated on a 7-point scale (1 = Extremely dissatisfied, 2=Very dissatisfied, 3=Somewhat dissatisfied, 4=Neither satisfied nor dissatisfied, 5=Somewhat satisfied, 6 = Very satisfied, 7 = Extremely satisfied).
Time Frame: Visit 5 (Week 8)
Population: Modified Intent-to-Treat (mITT) population (All patients who are enrolled and received KarXT through week 8) with available MSQ scores at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | KarXT
Number analyzed (Participants) | 2
Score on a scale | 6.00 (0.000)

ADVERSE EVENTS:
Time Frame: From first dose to 28 days post last dose (up to approximately 113 days)
Arm/Group | KarXT
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=4)
Schizophrenia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=4)
Dizziness (Nervous system disorders) | 1
Akathisia (Nervous system disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Abnormal dreams (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Post procedural hypothyroidism (Injury, poisoning and procedural complications) | 1
Nausea (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Red blood cells urine positive (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT05643170/Prot_SAP_000.pdf